CLINICAL TRIAL: NCT07247916
Title: Developing and Piloting an Implementation Strategy for a Brief, Motivational Interviewing-based Lethal Means Safety Counseling Intervention in Primary Care Settings
Acronym: CDA-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSR4-001-24W; 1IK2RD000503-01A2 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Suicide Prevention
Keywords: suicide; firearm; primary care; lethal means safety; motivational interviewing; self-injurious behavior
MeSH Terms: conditions — Suicide Prevention; Suicide; Self-Injurious Behavior | interventions — Architectural Accessibility

STUDY DESIGN:
Intervention Model Description: This pilot randomized controlled trial includes two arms: the experimental arm will have trained PCMHI clinicians deliver a brief motivational interviewing-based intervention to facilitate secure firearm storage; the control arm will have PCMHI clinicians review a suicide prevention pamphlet.
Who Masked: Outcomes Assessor
Masking Description: The research assistant (outcomes assessor) will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active control (Active Comparator): The control condition will entail a 5-minute review of a pamphlet on suicide prevention with the PCMHI clinician. This pamphlet is produced by the Veteran's Crisis Line and is widely available on the OSP suicide prevention website as a VHA resource. This condition will control for time and attention, subject matter, mode of delivery, and setting.
  Interventions: Behavioral: Active control
- RAMP (Experimental): Participants randomized to the intervention condition will receive a brief, motivational interviewing-based intervention called RAMP (Raise the subject, Assess current storage, Motivate change, and Plan next steps) in the context of their clinical care. RAMP incorporates evidence-informed intervention components to facilitate secure firearm storage
  Interventions: Behavioral: RAMP

INTERVENTIONS:
Behavioral: RAMP — Participants randomized to the intervention condition will receive a brief, motivational interviewing-based intervention called RAMP (Raise the subject, Assess current storage, Motivate change, and Plan next steps) in the context of their clinical care. RAMP incorporates evidence-informed intervention components to facilitate secure firearm storage
  Arms: RAMP
Behavioral: Active control — The control condition will entail a 5-minute review of a pamphlet on suicide prevention with the PCMHI clinician. This pamphlet is produced by the Veteran's Crisis Line and is widely available on the OSP suicide prevention website as a VHA resource. This condition will control for time and attention, subject matter, mode of delivery, and setting.
  Arms: Active control

SUMMARY:
Suicide prevention remains a significant priority and nearly three-quarters of Veteran suicides result from firearm injury. Since access to lethal means of self-harm increases the risk of injury, the VA/DoD Clinical Practice Guidelines recommend that Veterans with elevated suicide risk receive lethal means safety (LMS) counseling to reduce access to lethal means, including firearms. However, no LMS counseling interventions have been tested within VA. Thus, the aim of this study is to conduct a pilot randomized controlled trial to evaluate the feasibility and acceptability of a tailored LMS counseling intervention compared to an active control condition.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial of up to 50 Veterans to assess the feasibility and acceptability of a LMS intervention and testing procedures.

ELIGIBILITY:
Inclusion Criteria:

For Veterans:

* Has access to a firearm
* Referred to PCMHI care

For clinicians (delivering intervention):

* deliver care in PCMHI
* trained in RAMP and study procedures

Exclusion Criteria:

For Veterans:

* Unable to consent due to cognitive impairment, severity of illness (including psychiatric symptoms), intoxication with drugs and/or alcohol
* Unreliable telephone access
* Inability to read English or communicate in spoken and written English

For clinicians (delivering intervention):

- Did not participate in training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening | through study completion, approximately 2 years
  Investigators will assess the number of new PCMHI patients seen in PCMHI and the number who were approached about potential study participation per month
Recruitment | through study completion, approximately 2 years
  Investigators will track the number of eligible Veterans who enrolled in the study per month
Retention | approximately 30 days
  Investigators will calculate the number of Veterans who received RAMP who were willing to complete immediate and one-month follow up assessments.
Assessment of behavioral outcomes | approximately 30 days
  Investigators will assess the percentage of participants who completed behavioral outcome measures within the time allotted at each timepoint
Veteran acceptability - Theoretical Framework of Acceptability | At immediate follow up, within approximately 2 weeks of intervention
  Investigators will assess Veteran acceptability using the eight Likert-style items from the Theoretical Framework of Acceptability questionnaire, which assess seven component constructs of acceptability including Veteran's experience of the lethal means safety intervention. Each item has 5 answer options (1-5) on a Likert Scale. Score range is 8 to 40, with a higher score indicating more higher reported acceptability.
Veteran acceptability - Experience and Satisfaction with intervention | At immediate follow up, within approximately 2 weeks of intervention
  Investigators will conduct qualitative evaluation of the participant's experience and satisfaction receiving the intervention.
Clinician acceptability - Theoretical Framework of Acceptability | at 50% enrollment (approximately 1 year) and 100% enrollment (approximately 2 years)
  Investigators will invite clinicians to respond to the eight-item Theoretical Framework of Acceptability questionnaire eliciting clinician acceptability of the lethal means safety intervention. Each item has 5 answer options (1-5) on a Likert Scale. Score range is 8 to 40, with a higher score indicating more higher reported acceptability.
Clinician acceptability - Negative impact | at 50% enrollment (approximately 1 year) and 100% enrollment (approximately 2 years)
  Investigators will assess to what extent PCMHI clinicians agree that study recruitment negatively impacted clinical care, using Likert-type items where '1' indicates "strongly disagree" and '5' indicates "strongly agree." For those responding >3 ("don't know"), an open-ended question will elicit detailed information (e.g., interfered with delivery of clinical care, led to Veteran frustration).

CONTACTS AND LOCATIONS:
Overall Officials: Frances Aunon, PhD MS, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No